CLINICAL TRIAL: NCT02564003
Title: Oxycodone Pharmacokinetics in Preterms, Infants and Children
Brief Title: Oxycodone Pharmacokinetics in Preterm Infants
Acronym: oksineoinfa
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Collaborators: Admescope Ltd (Industry)
Responsible Party: Principal Investigator, Merja Kokki, MD, Docent, Kuopio University Hospital
Other Study IDs: 2011-11-11
Record Dates: First submitted 2015-09-25; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Oxycodone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and urine samples for oxycodone concentration measurement
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Oxycodone: Oxycodone 0,1 mg/kg iv
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — oxycodone 0,1 mg/kg iv

SUMMARY:
The pharmacokinetics of oxycodone is well characterized in children older than six months of age. However, only one study has been published with children younger than six months, concluding that unexplained inter-individual variability is pronounced in the youngest children. The aim of the current study was to quantify oxycodone pharmacokinetics in children ranging from preterm newborn infants to children up to two years of age.

ELIGIBILITY:
Inclusion Criteria:

* Infants scheduled for surgery with planned perioperative or postoperative opioid analgesia were screened if the gestational age (GA) was at least 23 weeks and postnatal age (PNA) below 2 years

Exclusion Criteria:

* He/she had allergy or hypersensitivity to oxycodone or other ingredients in the formulations or had received monoamineoxidase, CYP3A (cytochrome P450 3A enzymes) or CYP2D6 (cytochrome P450 2D6 enzyme) inhibitors during the previous month or other reason that was considered to contraindicate participation.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children age from 23 gestational weeks to two years
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2012-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration of oxycodone | time zero hours to 24 hours